CLINICAL TRIAL: NCT03440970
Title: Mechanism and Effects of Manipulating Chloride Homeostasis in Stable Heart Failure
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 2000022016; 1R01HL139629-01 (NIH)
Record Dates: First submitted 2018-02-14; First posted 2018-02-22 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Decompensated Heart Failure
Keywords: Chloride homeostasisH

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Lysine Chloride (Experimental): Patients will be randomized to receive either lysine chloride or placebo. Patients will receive the study drug thrice daily for 5 days of randomized therapy, starting after the completion of a blood volume assessment.
  Interventions: Drug: Lysine Chloride
- Placebo (Placebo Comparator): Patients will be randomized to receive either lysine chloride or placebo. Patients will receive the study drug thrice daily for 5 days of randomized therapy, starting after the completion of a blood volume assessment.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Lysine Chloride — Patients will receive the study drug thrice daily for 5 days.
  Arms: Lysine Chloride
Other: Placebo — Patients will receive the placebo thrice daily for 5 days.
  Arms: Placebo

SUMMARY:
This study is designed to investigate the quantitative effects of sodium-free chloride supplementation on electrolyte balance, volume status, and sodium avidity in stable heart failure patients in a highly controlled environment.

DETAILED DESCRIPTION:
The overarching goal of this study is to develop a comprehensive understanding of the biology and therapeutic potential of sodium-free chloride supplementation. While sodium homeostasis has been the focus of substantial investigation, very little research has been devoted to understanding chloride homeostasis. Thus, this proposal is designed to obtain the full spectrum of information pertaining to chloride, such as novel areas with great interest by the scientific community (i.e. modulation of the WNK-kinase system and the use of exosomes), to more practical/basic questions (i.e. what happens to sodium chloride balance when a patient is challenged with chloride).

This study is designed as a highly controlled inpatient "GCRC" arm to be compared to a real world efficacy study that has been proposed as a separate study. With extensive biobanking and analysis of samples in the inpatient setting, we will be able to deliver a great wealth of information on the biology and therapeutic potential of manipulating chloride homeostasis in heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Meticulous history of medical compliance and attendance of appointments
* Stable heart failure as defined by:

  1. Absence of hospitalizations for 90 days
  2. Stable diuretic and medical therapy for 30 days
  3. Opinion of the patient's treating physician (Heart Failure Cardiologist) that the patient is at optimal volume status
* Evidence based heart failure treatment with maximally-tolerated doses of a beta blocker, ACE/ARB/neprilysin inhibitor and aldosterone antagonist
* Chronic loop diuretic therapy with ≥ 40 mg of furosemide equivalents
* Serum chloride <102 mmol/L

Exclusion Criteria:

* Inability to commit to or comply with the rigorous study protocol
* Use of a thiazide diuretic in the last 30 days
* History of metabolic or respiratory acidosis
* Use of metformin, acetazolamide, or any other agent that could predispose to acidosis. Patients who are on metformin may be enrolled if their metformin can be safely discontinued for the randomized periods in each arm. Any participants who have consistently elevated Blood glucose readings > 200 mg/dL while inpatient will not be enrolled.
* Serum bicarbonate level <24mmol/L
* Serum pH <7.3
* Estimated glomerular filtration rate <30 mL/min or prior or current history of renal replacement therapy
* Anemia, as defined by Hemoglobin <8.0 g/dL at screening visit
* Urinary incontinence or significant bladder dysfunction (post-void residual at screening >300 mL)
* Use of chloride containing medications that provide more than 5 mmol/day of chloride if the medication cannot be discontinued or substituted
* Appears unlikely, or unable to participate in the required study procedures, as assessed by the study PI or research RN (ex: clinically-significant psychiatric, addictive, or neurological disease)
* Inability to give written informed consent or follow study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2025-08-30 (Actual); Study Completion 2025-08-30 (Actual)

PRIMARY OUTCOMES:
Change in Blood Volume | Daily for 7-days
  Volumex is albumin labeled with the iodine isotope I-131 and is an FDA-approved method used to determine total blood volume. A linear mixed effect model will be used to analyze the trial with class variables of time and treatment group. Daily measures of blood collection will be compared across the 7 day collection period between intervention and placebo arms.

SECONDARY OUTCOMES:
Change in Serum Creatinine | Daily for 7-days
  A linear mixed effect model will be used to analyze the trial with class variables of time and treatment group. Daily measures of serum creatinine will be compared across the 7 day collection period between intervention and placebo arms.
Change in Cystatin C | Daily for 7-days
  A linear mixed effect model will be used to analyze the trial with class variables of time and treatment group. Daily measures of cystatin C will be compared across the 7 day collection period between intervention and placebo arms.
Change in Chloride | Daily for 7-days
  A linear mixed effect model will be used to analyze the trial with class variables of time and treatment group. Daily measures of chloride will be compared across the 7 day collection period between intervention and placebo arms.
Change in Bicarbonate | Daily for 7-days
  A linear mixed effect model will be used to analyze the trial with class variables of time and treatment group. Daily measures of bicarbonate will be compared across the 7 day collection period between intervention and placebo arms.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey M Testani, MD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No